CLINICAL TRIAL: NCT03736291
Title: The Effect of Repetitive Transcranial Magnetic Stimulation in Schizophrenia--A Randomized , Double-blind fMRI Study
Brief Title: The Effect of Repetitive Transcranial Magnetic Stimulation in Schizophrenia
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: There are two reasons why the study was stopped. One is that the machine to opreate MRI was damaged and we could not fix it. The second reason is the main reasearch fellow has graduated and there is no one else to conitune this project.
Sponsor: Shanghai Mental Health Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: JunCai
Record Dates: First submitted 2018-11-06; First posted 2018-11-09 (Actual); Last update posted 2021-09-27 (Actual); Status verified 2021-09

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- active rTMS (Active Comparator): The Active rTMS: The magnetic head uses the Magro X100's "8"-shaped coil, and the intervention site is the cerebellar vermis (1 cm below the occipital carina). The stimulation intensity is gradually increased by the 80%-100% exercise threshold according to the patient's tolerance. The total number of stimulation pulses per day is 600, the basic frequency is 5 Hz, and one short burst stimulus is given every 200 milliseconds. In each short array, three single pulses with a frequency of 50 Hz are buried, and every 10 short bursts are stimulated for 8 s. A total of 200 short bursts of stimulation. Intervention once a day, 5 times a week, intervention for 2 weeks, a total of 10 times.
  Interventions: Device: Repetitive transcranial magnetic stimulation
- sham rTMS (Sham Comparator): The sham rTMS: The sham stimulation method was to invert the "8" shaped coil, which was 180° to the scalp, and other intervention parameters were consistent with the study group.
  Interventions: Device: Repetitive transcranial magnetic stimulation

INTERVENTIONS:
Device: Repetitive transcranial magnetic stimulation — Repetitive Transcranial Magnetic Stimulation (rTMS) is a widely used non-invasive neuromodulation technique that induces excitatory changes in the cerebral cortex stimulated by repeated pulsed magnetic fields on the scalp.

SUMMARY:
Repetitive Transcranial Magnetic Stimulation (rTMS) can modulate neuronal activity and has been shown to improve symptoms in patients with schizophrenia, but the underlying neural mechanism is unknown.This study hypothesized that repetitive transcranial magnetic stimulation of the cerebellar vermis can alter the ciliary-related functional connections in schizophrenia, thereby improving negative symptoms, cognitive function, and emotional symptoms. Therefore, this study will firstly explore the difference in cerebellar functional connectivity between patients and healthy controls, and on this basis, patients undergo a resting state functional magnetic resonance scan before and after rTMS intervention in the cerebellar vermis, and observe the cerebellar function connection in the treatment. Before and after changes, analyze the relationship between these changes and clinical efficacy to explore the neural mechanisms of efficacy.

DETAILED DESCRIPTION:
Repetitive Transcranial Magnetic Stimulation (rTMS) can modulate neuronal activity and has been shown to improve symptoms in patients with schizophrenia, but the underlying neural mechanism is unknown.This study hypothesized that repetitive transcranial magnetic stimulation of the cerebellar vermis can alter the ciliary-related functional connections in schizophrenia, thereby improving negative symptoms, cognitive function, and emotional symptoms. Therefore, this study will firstly explore the difference in cerebellar functional connectivity between patients and healthy controls, and on this basis, patients undergo a resting state functional magnetic resonance scan before and after rTMS intervention in the cerebellar vermis, and observe the cerebellar function connection in the treatment. Before and after changes, analyze the relationship between these changes and clinical efficacy to explore the neural mechanisms of efficacy.

1. Aim of the study 1.1 Using resting state functional magnetic resonance imaging to observe the differences in cerebellar functional connections between schizophrenia patients and healthy controls, and to further understand the role of cerebellar abnormalities in the clinical symptoms of schizophrenia; 1.2 Provide evidence-based evidence and imaging evidence for the clinical efficacy of rTMS intervention in cerebellar palsy for patients with schizophrenia, and further understand the neural mechanism of efficacy.
2. Content of the study 2.1 Based on previous studies, this study will use resting-state functional magnetic resonance imaging to observe abnormalities in behavioral and cerebellar neural networks in patients with schizophrenia compared with healthy controls, and to explore these abnormalities and schizophrenia. The relationship between clinical symptoms. 2.2 According to the research hypothesis, this study will perform a resting-state functional magnetic resonance scan of the patient before and after rTMS intervention in the cerebellar vermis. The functional connection analysis method is used to observe the changes of the cerebellar nerve network before and after treatment, and the imaging data and clinical evaluation. The data of the scale is combined to explore the neural mechanisms of treatment.
3. Study design This study used resting-state functional magnetic resonance imaging to investigate the differences in cerebrospinal function connections between schizophrenia and healthy controls. Based on this, a randomized double-blind control design was used to study the repetitive transcranial magnetic stimulation of the cerebellar vermis for patients with schizophrenia. The clinical efficacy of the treatment and the neural mechanisms of the therapeutic effect. Inpatients with schizophrenia were admitted to the Shanghai Mental Health Center, and patients who met the criteria and successfully enrolled were randomly grouped (by random number table method), corresponding to the rTMS true stimulation group or the rTMS pseudo-stimulation group. Except for the rTMS operator, neither the patient nor the evaluator of the scale knew the patient's grouping.

ELIGIBILITY:
Inclusion Criteria:

* The patient met the diagnostic criteria for schizophrenia in DSM-IV;
* 18-55 years old;
* Right handed;
* On stable doses of psychotropic medications.

Exclusion Criteria:

* DSM-IV diagnosis of other Axis I disorders；
* Contraindications to TMS or MRI；
* Patients receiving ECT (electro-convulsive therapy) in last 6months；
* Left-handedness。

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2019-12 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
FCS | 4 weeks
  FCS (functional connectivity strength) value. The Pearson's correlation analysis was used to analyze the time series signals of the brain voxels, and the functional connection matrix model of each subject was established. The gray matter template is used to calculate the mean value of the functional connection between each brain voxel and other voxels, which is the FCS value of the voxel.

SECONDARY OUTCOMES:
PANSS | 4 weeks
  The clinical efficacy was determined according to the PANSS reduction rate. The PANSS reduction rate was calculated as the difference between the PANSS total score before and after treatment divided by the pre-treatment PANSS total score. The PANSS reduction rate was judged to be significant progress, progress, and ineffective by 50% to 100%, 20% to 49%, and 0 to 19%, respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Jun Cai, Study Director — Shanghai Mental Health Center

IPD SHARING:
Plan to Share IPD: No